CLINICAL TRIAL: NCT03798873
Title: Examining the Impact of the Use of a Custom-fitted, FeelWell™ Compression Garment to Improve the Quality of Life of Individuals With a BMI ≥35
Brief Title: Impact of the Use of FeelWell™ Compression Garment on Individuals With a BMI ≥35
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Feelwell Compression (Industry)
Collaborators: Washington Center for Weight Management and Research, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FeelWell2018
Record Dates: First submitted 2018-12-13; First posted 2019-01-10 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Obesity, Abdominal; Mobility Limitation; Quality of Life; Back Pain; Pain, Chronic; Weight Change, Body; Inactivity; Exercise; Body Composition; Redundant Skin
Keywords: Compression garment; Physical therapy; Obesity; Movement; Abdominal binder
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Mobility Limitation; Back Pain; Chronic Pain; Body Weight Changes; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Test group treated with the FeelWell™ Compression garment and control group without compression garment. All subjects will receive the same intervention working with exercise physiologist and physical therapist in order to improve mobility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FeelWell™ Compression garment use with increase mobility (Experimental): Subjects are randomized to wear custom-fitted FeelWell™ Compression garment daily during regular and exercise activities.
  Subjects will work with physical therapist and exercise physiologist to increase strength, mobility and activity.
  Interventions: Device: FeelWell™ Compression garment; Behavioral: Increase Mobility
- Increase mobility (Other): For the control group, subjects will work with physical therapist and exercise physiologist to increase strength, mobility and activity. The control group will not be assigned a compression garment during the trial.
  Interventions: Behavioral: Increase Mobility

INTERVENTIONS:
Device: FeelWell™ Compression garment — Registered FDA class I device:
  The FeelWell™ Compression garment is a custom-made orthopedic abdominal binder with full or half-body support. The garments are made of 70% polyamide and 30% elastane and OEKO-TEX certified confirming human-ecological safety of textiles. The company uses a wrap knitting to ensure an optimal compression and durability. The garment has two 360 degrees whalebones in the front and two in the back to provide support for the posture, reinforcing compression on the abdomen and lower-back.
  Arms: FeelWell™ Compression garment use with increase mobility
Behavioral: Increase Mobility — Subjects will work with exercise physiologist and physical therapist to increase mobility, strength and activity

SUMMARY:
To assess the effect of wearing a custom-fitted, FDA-registered, Class I device, compression garment (Obesinov, S.A.R.L.) by an individual with a BMI ≥ 35 on his/her day-to-day quality of life over a period of one year. Various measures of quality of life will be taken, including assessing an individual's level of pain, mood, self-stigma and comfort with the use of a compression garment. Additionally, to assess the impact of the compression garment on activity, strength, posture and movement of an individual with a BMI ≥35 over the period of one year.

DETAILED DESCRIPTION:
Individuals suffering with obesity often experience daily pain and discomfort which limits movement, a critical factor in managing weight, cardio-metabolic health, mood, sleep, self-esteem and ultimately overall quality of life. Many individuals who experience weight gain have an abdominal or central distribution of weight which affects body mechanics leading to back pain, poor posture, difficulty walking with altered gait, knee, foot, ankle and leg pain (IT band, meralgia paresthetica) and other non-specific chronic pain. Chronic pain impedes mobility often incorporating depression and low motivation in an endless cycle. Furthermore, as individuals are losing weight, they often suffer from excess skin which also aggravates by chafing (arms, inner thighs), hanging down and interfering with gait.

The Investigators will examine the effect of wearing a custom-fitted, FDA-registered, Class I device, compression garment (Obesinov, S.A.R.L.) by participants with a BMI ≥ 35 on day-to-day quality of life over a period of one year. Various measures of quality of life will be taken, including assessing the participant's level of pain, mood, self-stigma and comfort with the use of a compression garment. Additional assessments include impact of the compression garment on activity, strength, posture and movement as well as potential impact of the use of this garment on weight loss and change in laboratory measures of metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, over 18 years old.
* Subjects with a BMI of ≥ 35.
* Subjects in any stage of weight loss or maintenance.

Exclusion Criteria:

* Inability to put on or have help in putting on garment.
* Inability to participate in movement and exercise intervention.
* Panniculus grade >3 at baseline or other body habitus that limits mobility.
* Duke Activity Status Index (DASI) score < 3.62
* Medical condition limiting participation in trial or basic mobility.
* Current participation in a physical therapy program.
* Unwillingness to participate fully in trial.
* Participation in another trial at the same time.
* Patient Health Questionnaire (PHQ)-9≥15.
* Current or expected pregnancy
* Investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
6- minute walk test- distance walked | baseline, 1, 3, 6 and 12 months
  6-min walk test is a sub-maximal exercise test measuring the total distance walked by a subject in a period of 6 minutes to assess functional capacity of a subject's cardio-respiratory systems and reflects their ability to perform Activities of Daily Living. Total distance walked will be measured and change recorded from baseline.
6- minute walk test- Perceived exertion | baseline, 1, 3, 6 and 12 months
  The Borg Rate of Perceived Exertion scale of 1-10 will be used for the subject to record their exertion level from 1 (no exertion)-10 (maximal exertion) and change will be noted from baseline.
SF-36 physical component sub-score | baseline, 3, 6 and 12 months
  SF-36 consists of 8 sub-scales of health-related quality of life measuring various aspects of functioning. The summary score for physical component includes physical functioning, physical role, bodily pain and general health scores. This sub-score is reported on a scale from 0-100 with higher numbers indicating better physical functioning.
30 Second Chair Stand | baseline, 1, 3, 6 and 12 months
  A test of leg strength and endurance. The number of times a patient stands from a sitting position in 30 seconds is recorded.
Brief Pain Inventory-Interference sub-score | baseline, 1, 3, 6 and 12 months
  A measure of pain and the interference of such pain on daily function. A sub-score on a scale of 0 (no interference)- 10 (maximal interference) will be recorded. The mean score of the 7 items will be recorded.
Steps per day measured by accelerometer | baseline, 6 months and 1 year
  The number of steps per day will be recorded as a measure of daily activity and averaged at various time points throughout the trial.
Weight Self Stigma questionnaire | baseline, 1, 3, 6 and 12 months
  A questionnaire designed to explore both internalized self stigma (internalized self-devaluation) and enacted stigma (directly experienced stigma) on function will be administered. The scale is comprised of 12 questions, and the subject responds on a scale from 1-5 with a greater score indicating greater experienced stigma.

SECONDARY OUTCOMES:
Lean body mass | baseline, 12 months
  Using DXA (Dual-energy X-ray Absorptiometry), lean body mass (LBM) or fat-free mass will be measured at baseline and at end of study. Percent change will be reported.
Fat mass | baseline, 12 months
  Using DXA (Dual-energy X-ray Absorptiometry), fat mass will be measured at baseline and at end of study. Percent change will be reported.
Bone density | baseline, 12 months
  Using DXA (Dual-energy X-ray Absorptiometry), bone density will be measured at baseline and at end of study. Percent change will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Domenica Rubino, MD, Principal Investigator — Washington Center for Weight Management and Research
Locations (1):
- Washington Center for Weight Management and Research, Inc., Shirlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Once study is completed, data analyzed and published, data will be made available to any investigator who is interested upon written request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of publication.
Access Criteria: Researchers must provide evidence that the data are being requested for analysis in a scientific study.

REFERENCES:
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Camarri B, Eastwood PR, Cecins NM, Thompson PJ, Jenkins S. Six minute walk distance in healthy subjects aged 55-75 years. Respir Med. 2006 Apr;100(4):658-65. doi: 10.1016/j.rmed.2005.08.003. Epub 2005 Oct 17. PMID 16229997
- [Background] Grodin JL, Hammadah M, Fan Y, Hazen SL, Tang WH. Prognostic value of estimating functional capacity with the use of the duke activity status index in stable patients with chronic heart failure. J Card Fail. 2015 Jan;21(1):44-50. doi: 10.1016/j.cardfail.2014.08.013. Epub 2014 Aug 28. PMID 25175697
- [Background] Jakicic JM, Rogers RJ, Davis KK, Collins KA. Role of Physical Activity and Exercise in Treating Patients with Overweight and Obesity. Clin Chem. 2018 Jan;64(1):99-107. doi: 10.1373/clinchem.2017.272443. Epub 2017 Nov 20. PMID 29158251
- [Background] Hebert-Losier K, Wessman C, Alricsson M, Svantesson U. Updated reliability and normative values for the standing heel-rise test in healthy adults. Physiotherapy. 2017 Dec;103(4):446-452. doi: 10.1016/j.physio.2017.03.002. Epub 2017 Mar 21. PMID 28886865